CLINICAL TRIAL: NCT00753129
Title: Influence of Head Elevation in Prone Position on Gas Exchange and Lung Mechanics in Patients With ALI/ARDS
Brief Title: Head Elevation in Prone Position
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Thomas Staudinger, MD, Dept. of Internal Medicine I, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EK 685/2007
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Gas Exchange; Lung Mechanics
Keywords: Prone position; ALI/ARDS; Head elevation
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Start with turning to prone position without head elevation, after 2 hours 30° head elevation, after 2 hours back to PP without head elevation.
  Interventions: Procedure: Prone position with head elevation
- 2 (Active Comparator): Start with turning to prone position with 30° head elevation, after 2 hours PP without head elevation, after 2 hours back to 0° PP.
  Interventions: Procedure: Prone position with head elevation

INTERVENTIONS:
Procedure: Prone position with head elevation — Head elevation of 30° in prone position (Ant-Trendelenburg position of the whole bed)

SUMMARY:
Semi-recumbent position leads to improvement of gas exchange and lung mechanics in patients suffering from ALI or ARDS. Prone positioning leads to similar effects. To date, no data on the combination of these two positioning measures exist. The investigators hypothesize that head elevation in prone position leads to improvement in gas exchange and lung mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated
* ALI or ARDS
* No contraindications for prone position

Exclusion Criteria:

* Patient < 18 or > 89 years old
* Pregnancy
* Elevated intracranial pressure
* PaO2/FiO2 - ratio < 60
* ECMO
* Open abdomen
* Instable spine
* Malignant arrhythmias
* Severe hemodynamic instability

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | Study period (5 hours on 2 consecutive days)

SECONDARY OUTCOMES:
PaCO2, Compliance (Chest wall, lung, respiratory system) | Study period (5 hours on 2 consecutive days)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Internal Medicine I, Intensive Care Unit, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Robak O, Schellongowski P, Bojic A, Laczika K, Locker GJ, Staudinger T. Short-term effects of combining upright and prone positions in patients with ARDS: a prospective randomized study. Crit Care. 2011;15(5):R230. doi: 10.1186/cc10471. Epub 2011 Sep 29. PMID 21955757